CLINICAL TRIAL: NCT02016937
Title: Effects of Different Anesthesia Protocols on Mother Lactation in The Postpartum Period
Brief Title: Mother Lactation in The Postpartum Period
Acronym: lactation
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, yavuz demiraran, Associated Professor, Duzce University
Other Study IDs: leylakutlucan; Duzce University (Other: Ethics committee of noninvasive clinical researches)
Record Dates: First submitted 2013-12-04; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Maternal-Fetal Relations
Keywords: Anesthesia , lactation, birth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- group g: general anesthesia, n: 21
- group S: spinal anesthesia, n: 21
- group E: epidural anesthesia, n: 21
- group V: vaginal birth, without anesthesia, n: 21

SUMMARY:
In our study we aimed to compare the lactation process by mothers who were undergoing elective Caesarian section under general anesthesia, spinal anesthesia, epidural anesthesia and normal vaginal birth.

DETAILED DESCRIPTION:
Patients were randomly divided into 4 groups: group G (general anesthesia for Caesarean section, n=21), group S (spinal anesthesia for Caesarean section, n=21), group E (epidural anesthesia for Caesarean section, n=21), group V (normal vaginal birth without anesthesia, n=21). Blood sample of 3 mililiters was taken from all patients 2,5 hours before procedure and oxytocin and prolactin levels in this blood samples were determined. No patient received premedication. Group G (general anesthesia for Caesarean section) received preoxygenation with 100% oxygen for 3-5 minutes before intubation. In order to let fetus minimally affected by the anesthetic agents, induction was performed after the disinfection and covering up of surgery area. Induction was performed with propofol (2 mg/ kg) and rocuronium (0,6 mg/kg). After onset of neuromuscular block, patients were intubated with compression maneuver of cricoid cartilage. Controlled ventilation was provided with anesthesia machine Datex Ohmeda S/5 Avance with tidal volume of 8-10 ml/kg, respiration frequency of 10-12 min. Anesthesia was maintained with oxygen (50%) , air (50%), sevoflurane of 1 MAC. When necessary rocuronium 0,15 mg/kg was administered. After delivery of the newborn, fentanyl 1-1,5 mcg/ kg was administered.

Patients in group S (spinal anesthesia for Caesarean section) received 750-1000 mL of 0,9% NaCI solution (10-15 mL/kg) as infusion in 20-30 minutes. Under strict aseptic precautions a 25G Quincke spinal needle was introduced into L3-L4 or L4-L5 intervertebral space in midline approach in sitting posture, and, after confirming free flow of CSF, predetermined 10-11 mg of drug solution (hypertonic bupivacaine 0,5%) was injected. We let the operation begin when sensory and motor blockade were verified. Oxygen of 100% (3 L. min) was administered throughout the operation via nasal cannula.

Patients in group E (epidural anesthesia for Caesarean section) received 750-1000 mL of 0,9% NaCI solution (10-15 mL/kg) as infusion in 20-30 minutes. We conducted epidural anesthesia with 18-gauge Tuohy needle at L3-L4 or L4-L5 epidural space by midline approach at sitting position. 3 -5 minutes after injection of 3 ml lidocaine as test-dose, when the patient has no sign of subarachnoid injection like prickling in lower extremities or of intravascular injection like nausea, vomiting, tachicardia, tinnitus, a 20-gauge epidural catheter was inserted to cephalad. We injected 10 ml of 0.5% bupivacaine via epidural catheter. We let the operation begin when sensory and motor blockade were verified. Oxygen of 100% (3 L. min) was administered throughout the operation via nasal cannula.

Patients in all 3 groups were monitorised in the operation room with a monitor of Datex-Ohmeda and electrocardiogram (ECG), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), peripheral oxygen saturation (SPO2) were recorded. Efedrin 5-10 mg and/or atropin 0,5 mg was administered when significant hypotension and bradicardia occurred. After delivery of the newborn 30 IU of oxytocin in a 1000cc solution of 0,9% NaCI was infused and if patient was not hypertensive, methylergonovine of 0,2 mg was administered intramuscular.

Patients in group V (spontaneous vaginal birth without anesthesia) were spectated by gynecologists in the Clinic of Gynecology and Obstetrics during the delivery. They received no anesthesia.

In all groups blood samples were taken at the 24th hour after delivery and oxytocin and prolactin levels were measured. Plasma of blood samples taken before and after delivery were stored at a temperature of -80°C. Prolactin levels were determined with chemiluminescense immunoassay technique Cobas e 601 (Roche® Diagnostics, Mannheim, Germany) using a commercial kit (Roche®). Oxytocin levels were determined with a commercial ELISA kit (Cusabio Biotech CO. Ltd). By all patients onset time of lactation was recorded.

ELIGIBILITY:
Inclusion Criteria:

* elective caesarian section
* normal vaginal delivery.
* between 18-40 years old
* risk of American society of anesthesiology grade-2

Exclusion criteria :

* Non-elective cases, plural pregnancies,
* Preterm pregnancies,
* Fetal anomalies,
* Retardation of fetal development,
* Newborns with birthweight under 2500 grams,
* Infants with risk of aspiration of meconium or amnios,
* Pathologies affecting acid-base balance,
* Diabetes mellitus,
* Hypertension,
* Antepartum hemorrhage,
* COPD (chronic obstructive pulmonary disease),
* Rhesus incompatibility,
* Obstetric complications like congenital malformations,
* History of malignant hypertermia,
* Morbid obesity, opioid sensitivity,
* Alcohol or drug addiction,
* Diseases of coronary arteria,
* Congestive heart failure,
* Serious anemia,
* History of liver or kidney diseases,
* Hypovolemia, hypotension,
* Systemic inflammatory response syndrome,
* Sepsis,
* History of allergic reactions to drugs used in the study,
* History of drugs affecting lactation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 84 patients were included. 63 of them were undergoing elective caesarian section and 21 patients had normal vaginal delivery in the Clinic of Gynecology and Obstetrics. All patients were between 18-40 years old and with the risk of ASA II.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
onset time of lactation of mothers | 24 h
  By all patients onset time of lactation was recorded postoperatively

SECONDARY OUTCOMES:
hormon levels | 24 h
  In all groups blood samples were taken at the 24th hour after delivery and oxytocin and prolactin levels were measured. Plasma of blood samples taken before and after delivery were stored at a temperature of -80°C. Prolactin levels were determined with chemiluminescense immunoassay technique Cobas e 601 (Roche® Diagnostics, Mannheim, Germany) using a commercial kit (Roche®). Oxytocin levels were determined with a commercial ELISA kit (Cusabio Biotech CO. Ltd).

OTHER OUTCOMES:
Apgar scores | 5 min
  Neonate APGAR Scores 1st and 5th minutes were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Demiraran, Study Director — Duzce University School of Medicine
Locations (1):
- Anesthesiology Department, Düzce, Turkey (Türkiye)

REFERENCES:
- [Result] Volmanen P, Valanne J, Alahuhta S. Breast-feeding problems after epidural analgesia for labour: a retrospective cohort study of pain, obstetrical procedures and breast-feeding practices. Int J Obstet Anesth. 2004 Jan;13(1):25-9. doi: 10.1016/S0959-289X(03)00104-3. PMID 15321436
- [Result] Baumgarder DJ, Muehl P, Fischer M, Pribbenow B. Effect of labor epidural anesthesia on breast-feeding of healthy full-term newborns delivered vaginally. J Am Board Fam Pract. 2003 Jan-Feb;16(1):7-13. doi: 10.3122/jabfm.16.1.7. PMID 12583645
- [Result] Uvnas-Moberg K, Widstrom AM, Werner S, Matthiesen AS, Winberg J. Oxytocin and prolactin levels in breast-feeding women. Correlation with milk yield and duration of breast-feeding. Acta Obstet Gynecol Scand. 1990;69(4):301-6. doi: 10.3109/00016349009036151. PMID 2244461
- See also: http://www.tip.duzce.edu.tr/ — http://www.duzce.edu.tr/